CLINICAL TRIAL: NCT04169971
Title: A Prospective Randomised Controlled Trial to Investigate the Effects of Intra-operative Music on Anxiety Levels During Procedures Under Spinal Anaesthesia at a Surgical Centre in Cambodia
Brief Title: Investigation of the Effects of Music on Anxiety During Operations Under Spinal Anaesthesia at an Hospital in Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Surgical Center, Cambodia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: musicduringspinal1
Record Dates: First submitted 2019-10-31; First posted 2019-11-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-11

CONDITIONS: Surgery; Anxiety
Keywords: trial; Anxiety; music; intraoperative period; spinal anaesthesia
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: This is a single-centre, prospective, randomised controlled trial. Patients will be invited to participate if they are due to undergo a procedure for which they will require spinal anaesthesia and if they meet the inclusion criteria and none of the exclusion criteria. They will not be required to make any additional hospital visits and will be asked to give their informed consent prior to the procedure. Half of the participants will receive music from the start of surgery until completion of the operation and the other half will serve as the 'control group' and will receive no headphones or music. The anxiety of participant's during the operation will be assessed through a VAS and they will be asked questions about their experience afterwards. The anxiety scores from the two groups will be compared, as will their responses to the questions about their experience, in order to elucidate whether the music produced any differences in anxiety or experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): Will receive music during the operation conducted under spinal anaesthesia
  Interventions: Other: Music
- Control group (No Intervention): Will not receive music during the operation conducted under spinal anaesthesia

INTERVENTIONS:
Other: Music — Played through headphones during the operation under spinal anaesthesia
  Arms: Music group

SUMMARY:
This study investigates he effects of intra-operative music on anxiety levels during procedures under spinal anaesthesia at a surgical centre in Cambodia. Participants will be randomly allocated to either the music (M) group or the 'control' (C) group. The M group will receive music played through headphones for the duration of the operation. The C group will receive no music or headphones. Anxiety will be measured in both groups, through a visual analogue scale (VAS), at the beginning of the operation and after 30 minutes of the procedure. Scores will be compared.

DETAILED DESCRIPTION:
Background: During operations conducted under spinal anaesthesia patients are aware of their environment, including sounds related to operative instruments and the voices of staff. This has the potential to cause anxiety and amplify existing anxiety which can negatively impact patient experience and outcomes. Research has shown peri-operative music can reduce anxiety but there is no robust evidence for the effect of intraoperative music on intraoperative anxiety.

Objectives: The primary objective is to determine the effects of intraoperative music on intraoperative anxiety levels for patients undergoing procedures conducted under spinal anaesthesia. The secondary objectives are to investigate whether participants feel that music improved/would improve their experience and whether they would choose it in future or recommend it for others.

Methods: This prospective randomised controlled trial will be conducted at the Children's Surgical Centre in Phnom Penh. Participants will be 18 years or over, due to undergo a procedure that requires spinal anaesthesia and not have a medical history that fulfils any of the exclusion criteria. The trial will aim to recruit between 16 and 28 patients consecutively once it commences, and participants will be randomised to either the music (M) group or the 'control' (C) group. The M group will receive music (pre-selected from 5 categories) played through headphones for the duration of the operation. The C group will receive no music or headphones. Anxiety will be measured in both groups, through a visual analogue scale (VAS), at the beginning of the operation and after 30 minutes of the procedure. In the recovery room the participants will be asked two questions relating to experience and future recommendations.

Results: The VAS scores and change in VAS scores will be displayed as mean ± Standard Error and the results from the two groups will be compared using a student's paired t-test or a Mann-Whitney U test depending on the distribution of the data. The results from the post-operation questions will be displayed as frequencies and the answers will be compared using a χ2 test. All tests will be 2-tailed and P<0.05 will be considered significant

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Undergoing a procedure at CSC that requires spinal anaesthesia and spinal anaesthesia is not contra-indicated
* Gives informed consent to participate in the trial

Exclusion Criteria:

* Has an existing psychological diagnosis
* Has auditory impairment
* Deemed not to have capacity to give consent
* Sedatives are administered during the procedure
* General anaesthesia is required during the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Change in intra-operative anxiety scores | Calculated between scores recorded at the start of the operation and 30 minutes into the procedure
  Score on 'Anxiety visual analogue scale.' Minimum score 0 representing calm and maximum score 10 representing extreme anxiety

SECONDARY OUTCOMES:
Percentage of patient's in the music group who felt that music made the experience better, worse or had no effect. | Within 4 hours post operation
  Questionnaire asked verbally. What effect do you think music had on your experience during surgery? a) made it better b)made it worse c)no effect.
Percentage of patient's in the music group who felt that they would recommend to others, wouldn't recommend to others or did not know. | Within 4 hours post operation
  Questionnaire asked verbally. Would you recommend listening to music during an operation to other people? a)yes b)no c) don't know
Percentage of patient's in the control group who felt that music would have made their experience better, worse or the same. | Within 4 hours post operation
  What effect do you think music would have had on your experience during surgery? a) made it better b)made it worse c)no effect.
Percentage of patient's in the music group who, if they had another operation, would like to listen to music, would not like to listen to music, or did not know. | Within 4 hours post operation
  Questionnaire asked verbally. Would you like to listen to music if you were to have another operation? a)yes b)no c) don't know
Percentage of anaesthetic providers that experience problems due to music. | Within 4 hours post operation
  Questionnaire on data collection form. Do you think that the music caused any problems during the operation? a)yes b)no c)maybe

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Larvin, BMBCH, Principal Investigator — Children's Surgical Centre, Phnom Penh, Cambodia; SOKHALAY L SUOS, MD, Principal Investigator — Children's Surgical Centre, Phnom Penh, Cambodia
Locations (1):
- Children's Surgical Centre, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after recruitment of last participant.
Access Criteria: Requests will be reviewed by an independent review panel and all requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Norris W, Baird WL. Pre-operative anxiety: a study of the incidence and aetiology. Br J Anaesth. 1967 Jun;39(6):503-9. doi: 10.1093/bja/39.6.503. No abstract available. PMID 6027959
- [Background] Caumo W, Schmidt AP, Schneider CN, Bergmann J, Iwamoto CW, Adamatti LC, Bandeira D, Ferreira MB. Risk factors for postoperative anxiety in adults. Anaesthesia. 2001 Aug;56(8):720-8. doi: 10.1046/j.1365-2044.2001.01842.x. PMID 11493233
- [Background] Wilson CJ, Mitchelson AJ, Tzeng TH, El-Othmani MM, Saleh J, Vasdev S, LaMontagne HJ, Saleh KJ. Caring for the surgically anxious patient: a review of the interventions and a guide to optimizing surgical outcomes. Am J Surg. 2016 Jul;212(1):151-9. doi: 10.1016/j.amjsurg.2015.03.023. Epub 2015 Jun 2. PMID 26138522
- [Background] Jlala HA, Bedforth NM, Hardman JG. Anesthesiologists' perception of patients' anxiety under regional anesthesia. Local Reg Anesth. 2010;3:65-71. doi: 10.2147/lra.s11271. Epub 2010 Aug 12. PMID 22915871
- [Background] Wu PY, Huang ML, Lee WP, Wang C, Shih WM. Effects of music listening on anxiety and physiological responses in patients undergoing awake craniotomy. Complement Ther Med. 2017 Jun;32:56-60. doi: 10.1016/j.ctim.2017.03.007. Epub 2017 Mar 31. PMID 28619305
- [Background] Zengin S, Kabul S, Al B, Sarcan E, Dogan M, Yildirim C. Effects of music therapy on pain and anxiety in patients undergoing port catheter placement procedure. Complement Ther Med. 2013 Dec;21(6):689-96. doi: 10.1016/j.ctim.2013.08.017. Epub 2013 Sep 1. PMID 24280479
- [Background] Costa A, Montalbano LM, Orlando A, Ingoglia C, Linea C, Giunta M, Mancuso A, Mocciaro F, Bellingardo R, Tine F, D'Amico G. Music for colonoscopy: A single-blind randomized controlled trial. Dig Liver Dis. 2010 Dec;42(12):871-6. doi: 10.1016/j.dld.2010.03.016. Epub 2010 May 7. PMID 20452299
- [Background] Pittman S, Kridli S. Music intervention and preoperative anxiety: an integrative review. Int Nurs Rev. 2011 Jun;58(2):157-63. doi: 10.1111/j.1466-7657.2011.00888.x. Epub 2011 Feb 15. PMID 21554287
- [Background] Tan X, Yowler CJ, Super DM, Fratianne RB. The efficacy of music therapy protocols for decreasing pain, anxiety, and muscle tension levels during burn dressing changes: a prospective randomized crossover trial. J Burn Care Res. 2010 Jul-Aug;31(4):590-7. doi: 10.1097/BCR.0b013e3181e4d71b. PMID 20498613
- [Background] Wang SM, Kulkarni L, Dolev J, Kain ZN. Music and preoperative anxiety: a randomized, controlled study. Anesth Analg. 2002 Jun;94(6):1489-94, table of contents. doi: 10.1097/00000539-200206000-00021. PMID 12032013
- [Background] McClurkin SL, Smith CD. The Duration of Self-Selected Music Needed to Reduce Preoperative Anxiety. J Perianesth Nurs. 2016 Jun;31(3):196-208. doi: 10.1016/j.jopan.2014.05.017. Epub 2016 Feb 24. PMID 27235956
- [Background] Mingir T, Ervatan Z, Turgut N. Spinal Anaesthesia and Perioperative Anxiety. Turk J Anaesthesiol Reanim. 2014 Aug;42(4):190-5. doi: 10.5152/TJAR.2014.99705. Epub 2014 May 29. PMID 27366419
- [Background] Lee WP, Wu PY, Lee MY, Ho LH, Shih WM. Music listening alleviates anxiety and physiological responses in patients receiving spinal anesthesia. Complement Ther Med. 2017 Apr;31:8-13. doi: 10.1016/j.ctim.2016.12.006. Epub 2017 Jan 7. PMID 28434475
- [Background] Lepage C, Drolet P, Girard M, Grenier Y, DeGagne R. Music decreases sedative requirements during spinal anesthesia. Anesth Analg. 2001 Oct;93(4):912-6. doi: 10.1097/00000539-200110000-00022. PMID 11574356
- [Background] Maeyama A, Kodaka M, Miyao H. [Effect of the music-therapy under spinal anesthesia]. Masui. 2009 Jun;58(6):684-91. Japanese. PMID 19522258
- [Background] Elkins G, Staniunas R, Rajab MH, Marcus J, Snyder T. Use of a numeric visual analog anxiety scale among patients undergoing colorectal surgery. Clin Nurs Res. 2004 Aug;13(3):237-44. doi: 10.1177/1054773803262222. PMID 15245638
- [Background] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Background] Seponski DM, Lahar CJ, Khann S, Kao S, Schunert T. Four decades following the Khmer rouge: sociodemographic factors impacting depression, anxiety and PTSD in Cambodia. J Ment Health. 2019 Apr;28(2):175-180. doi: 10.1080/09638237.2018.1466039. Epub 2018 May 7. PMID 29733242
- [Background] Alfredsson M, San Sebastian M, Jeghannathan B. Attitudes towards mental health and the integration of mental health services into primary health care: a cross-sectional survey among health-care workers in Lvea Em District, Cambodia. Glob Health Action. 2017;10(1):1331579. doi: 10.1080/16549716.2017.1331579. PMID 29261452